CLINICAL TRIAL: NCT00303212
Title: A Study of Telemonitoring to Improve Heart Failure Outcomes
Brief Title: Tele-HF: Yale Heart Failure Telemonitoring Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Harlan Krumholz. MD, Yale School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0502027466; R01HL080228 (NIH)
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2010-09

CONDITIONS: Congestive Heart Failure
Keywords: heart failure; CHF; telemedicine; disease management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UC (No Intervention): Usual HF guideline-base care
- TM (Experimental): Telemonitoring group plus usual guideline-based HF care
  Interventions: Other: Telemonitoring

INTERVENTIONS:
Other: Telemonitoring — Participants in the intervention group are instructed to make a daily toll-free call to an automated telemonitoring system being provided by Pharos Innovations® (Chicago, IL) for 6 months.On each call patients hear a pre-recorded voice that goes through a series of questions about symptoms and the patient's daily weight. Information from the telemonitoring system is automatically downloaded to a secure Internet site for review by clinicians at each practice site.
  Other Names: Tel-Assurance
  Arms: TM

SUMMARY:
The primary purpose of this study is to determine the effectiveness of telemonitoring compared with usual guideline-based care in preventing hospitalization for heart failure patients.

DETAILED DESCRIPTION:
Heart failure (HF) is a common, costly condition characterized by recurrent periods of clinical decompensation that often lead to repeated hospitalizations (1, 2). Despite advances in the care of patients with HF, population-based outcomes such as mortality and hospitalization rates have not improved substantially over the past decade (3). Episodic, infrequent, outpatient visits are the only usual opportunities for clinicians to detect and treat early signs of HF decompensation; this constitutes a major gap in the current medical model. Moreover, opportunities for patients to take an active role in managing their own conditions occur infrequently. Disease management has emerged as a possible solution to the need for better patient surveillance and engagement. It typically involves multidisciplinary efforts to improve the quality and efficiency of care for patients with chronic conditions, with interventions designed to foster adherence of clinicians to scientific guidelines and patients to treatment plans. However, traditional disease-management programs are generally resource-intensive (often relying on nurse case management), difficult to scale for a large population, and inefficient in providing daily patient monitoring.

Telemonitoring, which bridges clinicians and patients with communication technology, holds promise for closing the gap in HF care (4). This technology has the potential for standardized, widespread implementation (and long-term maintenance) in the near future because it can be easily applied to large patient populations and integrated into the current medical care system. Supporting this potential, preliminary evaluations have suggested that telemonitoring is feasible across a broad spectrum of typical HF patients, relatively inexpensive on a per-patient basis, and highly effective in improving health outcomes. Thus, this approach is ready for rigorous evaluation.

Accordingly, we propose an office-based, multicenter, randomized controlled trial (Tele-HF study) to determine the effectiveness of a telemonitoring strategy in decreasing hospital readmissions and death in patients with HF. Many HF patients experience deterioration in their health status and an increase in weight and symptoms over a period of days and weeks before ultimately presenting to medical attention and requiring hospitalization. Our premise is that a frequent monitoring system can alert clinicians to the early signs and symptoms of decompensation, providing the opportunity for intervention before the patient becomes severely ill and requires hospitalization. Moreover, such a system can engage patients in their care and provide instruction about beneficial self-care strategies. This intervention is not intended to substitute for communication relating to acute care or acute, sudden changes in health status. In these cases, patients are instructed to make direct and immediate contact with their doctor or hospital.

We will use the Pharos Tel-AssuranceTM, an in-home communication system that allows patients to transmit information to their clinicians and provides education to enable patients to actively participate in managing their condition. The system uses conventional telephone lines and does not require the patient to have Internet access. Patients are asked a pre-programmed series of questions and the system automatically uploads the responses to a secure data center. A clinician in each practice can then log on to a secure Internet site using a Web browser to review the patients' responses. The system thus serves as an interface between patients at home and their clinicians, facilitating monitoring of chronic conditions and patient education. While many vendors have potential tools to implement this study, we chose to use Pharos Tel-AssuranceTM because it is simple to use, does not require any equipment in patients' homes and substantial preliminary data suggest high patient and clinician satisfaction with its use. The investigators have no financial interest in this company.

Primary Aim Our primary aim is to determine whether telemonitoring by community-based cardiology office practices reduces the risk of hospital readmission (for any cause) or death after an initial "index hospitalization" for HF. We hypothesize that, among patients recently discharged after a hospitalization for HF, telemonitoring will decrease the rate of rehospitalization or death over 6 months by at least 15% (relative risk reduction). This would yield an absolute risk reduction of 7.5%, so that 1 major adverse event would be averted for every 13 patients.

We have chosen all-cause readmission as part of our primary outcome because poorly controlled HF can result in admissions for a variety of reasons, as the patient becomes weak and susceptible to falls, mental status changes, renal dysfunction, and other debilitating conditions that can result in hospitalization. In addition, from a societal and health system perspective, the overall risk of readmission is more important than disease-specific readmission. Moreover, prior studies suggest that telemonitoring can reduce this outcome.

Secondary Aims

In our secondary aims we will determine whether telemonitoring will:

1. Reduce the rate of all-cause hospital readmission
2. Reduce the rate of hospital readmission for HF
3. Reduce the total number of all-cause and HF-specific hospital readmissions
4. Increase office visits with the clinician receiving information from the telemonitoring system
5. Improve survival after index hospitalization
6. Reduce the cost of inpatient medical care
7. Improve health status
8. Improve patient satisfaction with care
9. Improve patients' self-management of HF

Sub-Group Analyses

The following sub-group analyses will be conducted:

1. Age
2. Sex
3. Race
4. HFPEF vs depressed EF
5. Education
6. Insurance status
7. Self-reported access to care
8. Baseline self-efficacy and self-care
9. Socioeconomic Status
10. Site characteristics

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* hospitalized for heart failure within the past 30 days
* access to telephone line

Exclusion Criteria:

* not expected to survive 6 months due to irreversible, life-threatening condition
* has or scheduled for cardiac transplant or LVAD
* scheduled for CABG or PCI within 90 days
* severe valvular disease
* Folstein MMSE score less than 20
* resident of a nursing home
* currently a prisoner
* does not speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1660 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Rate of all-cause hospital readmission or death during the 6-month follow-up period. | 6 months

SECONDARY OUTCOMES:
Rate of all-cause hospital readmissions | 6 months
Number of office visits with clinician receiving information from the telemonitoring system | 6 months
Survival after index hospitalization | 6 months
Cost of inpatient medical care | 6 months
Health status | 6 months
Patient satisfaction with care | 6 months
Patients' self-management of heart failure | 6 months
Post index discharge hospital days | 6 months
Post index discharge hospital days/follow up days alive | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Harlan M. Krumholz, M.D., Principal Investigator — Yale University; Sarwat I Chaudhry, MD, Study Director — Yale University; Jennifer Mattera, MPH, Study Director — Yale University
Locations (33):
- United States (33):
  - Cardiology Associates, Mobile, Alabama
  - UC Irvine Medical Center, Orange, California
  - UCLA Harbor Medical Center, Torrance, California
  - Department of Cardiology at Bridgeport Hospital, Bridgeport, Connecticut
  - Cardiology Associates of New Haven, New Haven, Connecticut
  - Howard University Hospital, Washington D.C., District of Columbia
  - Integrated Care / Cardiovascular Consultants of South Florida, Tamarac, Florida
  - Piedmont Hospital Research Institute, Atlanta, Georgia
  - Morehouse School of Medicine/Cardiology, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana Heart Physicians, Indianapolis, Indiana
  - Iowa City Heart Center, Iowa City, Iowa
  - Chabert Medical Center, Houma, Louisiana
  - Heart Clinic of Louisiana, Marrero, Louisiana
  - Cardiology Associates, LLC, Tupelo, Mississippi
  - Truman Medical Center/Cardiology, Kansas City, Missouri
  - St. Luke's Hospital / Mid-America Heart Institute, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Cardiology Diagnostics, St Louis, Missouri
  - Cooper Health System Cardiology, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - St. Joseph's Regional Medical Center / Cardiology Associates, Paterson, New Jersey
  - New York University/Cardiology, New York, New York
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Heart & Vascular Center, Cleveland, Ohio
  - The Dayton Heart Center, Dayton, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Cardiology Specialists, Ltd., Westerly, Rhode Island
  - Baylor University Medical Center, Dallas, Texas
  - Sentara Cardiology Consultants, Ltd., Norfolk, Virginia

REFERENCES:
- [Derived] Jayaram NM, Khariton Y, Krumholz HM, Chaudhry SI, Mattera J, Tang F, Herrin J, Hodshon B, Spertus JA. Impact of Telemonitoring on Health Status. Circ Cardiovasc Qual Outcomes. 2017 Dec;10(12):e004148. doi: 10.1161/CIRCOUTCOMES.117.004148. PMID 29237746
- [Derived] Steventon A, Chaudhry SI, Lin Z, Mattera JA, Krumholz HM. Assessing the reliability of self-reported weight for the management of heart failure: application of fraud detection methods to a randomised trial of telemonitoring. BMC Med Inform Decis Mak. 2017 Apr 18;17(1):43. doi: 10.1186/s12911-017-0426-4. PMID 28420352
- [Derived] Mortazavi BJ, Downing NS, Bucholz EM, Dharmarajan K, Manhapra A, Li SX, Negahban SN, Krumholz HM. Analysis of Machine Learning Techniques for Heart Failure Readmissions. Circ Cardiovasc Qual Outcomes. 2016 Nov;9(6):629-640. doi: 10.1161/CIRCOUTCOMES.116.003039. Epub 2016 Nov 8. PMID 28263938
- [Derived] Krumholz HM, Chaudhry SI, Spertus JA, Mattera JA, Hodshon B, Herrin J. Do Non-Clinical Factors Improve Prediction of Readmission Risk?: Results From the Tele-HF Study. JACC Heart Fail. 2016 Jan;4(1):12-20. doi: 10.1016/j.jchf.2015.07.017. Epub 2015 Dec 2. PMID 26656140
- [Derived] Qian F, Parzynski CS, Chaudhry SI, Hannan EL, Shaw BA, Spertus JA, Krumholz HM. Racial Differences in Heart Failure Outcomes: Evidence From the Tele-HF Trial (Telemonitoring to Improve Heart Failure Outcomes). JACC Heart Fail. 2015 Jul;3(7):531-538. doi: 10.1016/j.jchf.2015.03.005. PMID 26160368
- [Derived] Bikdeli B, Wayda B, Bao H, Ross JS, Xu X, Chaudhry SI, Spertus JA, Bernheim SM, Lindenauer PK, Krumholz HM. Place of residence and outcomes of patients with heart failure: analysis from the telemonitoring to improve heart failure outcomes trial. Circ Cardiovasc Qual Outcomes. 2014 Sep;7(5):749-56. doi: 10.1161/CIRCOUTCOMES.113.000911. Epub 2014 Jul 29. PMID 25074375
- [Derived] Chaudhry SI, Mattera JA, Curtis JP, Spertus JA, Herrin J, Lin Z, Phillips CO, Hodshon BV, Cooper LS, Krumholz HM. Telemonitoring in patients with heart failure. N Engl J Med. 2010 Dec 9;363(24):2301-9. doi: 10.1056/NEJMoa1010029. Epub 2010 Nov 16. PMID 21080835